CLINICAL TRIAL: NCT02207101
Title: The Effect of Investigational Product E-OJ-01 (OXYJUN) on Left Ventricular Ejection Fraction and Markers of Cardiovascular Injury.
Brief Title: Study to Assess the Effect of OXYJUN on Ejection Fraction and Markers of Cardiovascular Injury
Acronym: Enduoxy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Collaborators: Enovate Biolife Pvt Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: EB/141005/OXY-2/CE
Record Dates: First submitted 2014-07-21; First posted 2014-08-01 (Estimated); Last update posted 2015-07-10 (Estimated); Status verified 2015-07

CONDITIONS: Cardiac Function in Young Athletes
Keywords: Young athletes; Cardiac endurance; Herbal; Ejection Fraction; Basic Research; Cardiovascular Injury

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- E-OJ-01 (OXYJUN) (Active Comparator): E-OJ-01 (OXYJUN). Dose: 01 capsule to be taken orally daily after lunch.
  Interventions: Dietary Supplement: E-OJ-01 (OXYJUN)
- Placebo (Placebo Comparator): Matching placebo capsules [for E-OJ-01 (OXYJUN)] composed of microcrystalline cellulose. Dose: 01 capsule to be taken orally daily after lunch.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: E-OJ-01 (OXYJUN)
  Arms: E-OJ-01 (OXYJUN)
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
Young athletes are usually regarded as a special subgroup of healthy individuals with a unique lifestyle who are apparently invulnerable and often capable of extraordinary physical achievement. Most athletic disciplines to some extent combine endurance and strength modes of physical conditioning. Acute responses to endurance exercise training include substantial increases in maximal oxygen uptake, cardiac output, stroke volume, and systolic blood pressure in-spite of this, high intensity chronic training such as marathons, very long distance bicycle racing etc., can lead to transient acute volume overload of the atria and right ventricle, with transient reductions in right ventricular ejection fraction and elevations of cardiac biomarkers. Although these biomarkers generally normalize back within seven to ten days, these transient changes may sooner or later mark the beginning of processes like patchy myocardial fibrosis finally leading to grave chronic heart diseases .

Inspite of the awareness regarding the cardio vascular risk in the athletes, there have been no new advancements in finding an alternate option which can protect the cardio vascular system in the athletes.

Hence in order to address the need of the hour and also to avoid the cardio vascular risk in athletes along with improvising the endurance capacity, Enovate Biolife is in the process of development of an innovative product "E-OJ-01".

E-OJ-01 is expected to have beneficial effects on the cardio vascular system of the athletes by enhancing ejection fraction which in turn improves cardiac output. This finally is hypothysed to increase the maximal oxygen uptake capacity in athletes.

ELIGIBILITY:
Inclusion Criteria:

* Male athletes aged 18 - 40 years having endurance exercise not less than 3-4 hrs. / week since at least last 12 weeks.
* Subject with left ventricular ejection fraction not less than 55% and not more than 70%.
* Subjects having body fat less than 16% as determined by skin fold assessment.
* Subject is willing to refrain from vigorous physical activity 12 hrs prior to clinic visit.
* Subject is a non-alcoholic/ non-smoker.
* Subject understands the study procedures and signs forms providing informed consent to participate in the study and authorization for release of relevant protected health information to the study Investigator.

Exclusion Criteria:

* Left Ventricular Ejection fraction less than 55 per cent by echocardiogram.
* Subjects suffering from anemia as defined by Hb levels ≤ 10 g/ dl.
* Subject has uncontrolled hypertension (systolic blood pressure ≥160 mm Hg or diastolic blood pressure ≥ 100 mm Hg) as defined by the average blood pressure measured at screening.
* History of coronary artery disease, myocardial infarction, hypertension or diabetes mellitus.
* History of cardiomyopathy, congenital heart defect, open heart surgery, or ongoing arrhythmia.
* Subjects having laboratory finding beyond specified normal limits at screening and in the opinion of the investigator possess significant threat for the study subject.
* Subject has a history or presence of clinically important renal, hepatic, endocrine (including diabetes mellitus), pulmonary, biliary, gastrointestinal, pancreatic, or neurologic disorders that, in the judgment of the Investigator, would interfere with the subject's ability to provide informed consent, comply with the study protocol (which might confound the interpretation of the study results), or put the subject at undue risk.
* Use of any sleep aid medication within four days prior to each test day.
* Use of any psychotropic medication within four weeks of screening and throughout the study.
* Subject has a history, in the judgment of the Investigator, of a psychological illness or condition such as to interfere with the subject's ability to understand the requirements of the study.
* Use of antibiotics or signs of active systemic infection. Treatment visits will be rescheduled to allow the subject to wash off of the antibiotic for at least five days prior to any test visit. Use of any other dietary supplements or herbal products.
* Recent history of (within 12 months of screening visit 1) or strong potential for alcohol or substance abuse.
* Subject has a known allergy or sensitivity to herbal product(s).
* Subject has had exposure to any non-registered drug product within 30 days prior to the screening visit.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2014-12; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change in Left Ventricular Ejection Fraction | Day 0, Day 28 and Day 56

SECONDARY OUTCOMES:
Change in Serum Troponin-T | Day 0 and Day 56

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Chavan, MD, Principal Investigator
Locations (1):
- Suburban Diagnostics, Mumbai, Maharashtra, India

REFERENCES:
- [Derived] Girandola RN, Srivastava S. Effect of E-OJ-01 on Cardiac Conditioning in Young Exercising Adults: A Randomized Controlled Trial. Am J Ther. 2017 May;24(3):e298-e307. doi: 10.1097/MJT.0000000000000542. PMID 27930383